CLINICAL TRIAL: NCT02299089
Title: A Phase II, Open-label, Multicentre, Randomised Study of the Pharmacokinetics, Pharmacodynamics, Efficacy, and Safety of CAM2029 in Patients With Acromegaly and Neuroendocrine Tumours (NETs) Previously Treated With Sandostatin® LAR®
Brief Title: Phase II Study of Subcutaneous Inj. Depot of Octreotide in Patients With Acromegaly and Neuroendocrine Tumours (NETs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Camurus AB (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-12-455
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Acromegaly; Neuroendocrine Tumors
Keywords: acromegaly; neuroendocrine tumour (NET); carcinoid syndrome; octreotide; Sandostatin LAR
MeSH Terms: conditions — Acromegaly; Neuroendocrine Tumors; Serotonin Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CAM2029 10 mg (NET) (Experimental): CAM2029 (octreotide FluidCrystal® injection depot) 10 mg, subcutaneous injection every two weeks
  Interventions: Drug: octreotide FluidCrystal® injection depot
- CAM2029 20 mg (NET) (Experimental): CAM2029 (octreotide FluidCrystal® injection depot) 20 mg, subcutaneous injection once monthly
  Interventions: Drug: octreotide FluidCrystal® injection depot
- CAM2029 10 mg (Acromegaly) (Experimental): CAM2029 (octreotide FluidCrystal® injection depot) 10 mg, subcutaneous injection every two weeks
  Interventions: Drug: octreotide FluidCrystal® injection depot
- CAM2029 20 mg (Acromegaly) (Experimental): CAM2029 (octreotide FluidCrystal® injection depot) 20 mg, subcutaneous injection once monthly
  Interventions: Drug: octreotide FluidCrystal® injection depot

INTERVENTIONS:
Drug: octreotide FluidCrystal® injection depot
  Other Names: CAM2029

SUMMARY:
This is a Phase II, open-label multicentre, randomised study to assess the PK, PD, efficacy, and safety of two dosing regimens of CAM2029 in adult patients with acromegaly or a functional, well-differentiated NET, with carcinoid symptoms.

DETAILED DESCRIPTION:
This is a Phase II, open-label multicentre, randomised study to assess the PK, PD, efficacy, and safety of two dosing regimens of CAM2029 in adult patients with acromegaly or a functional, well-differentiated NET, with carcinoid symptoms, treated for at least 2 months with Sandostatin LAR at doses of 10 mg, 20 mg, or 30 mg before the start of the Sandostatin LAR Last Dose Assessment Phase (Day -28).

ELIGIBILITY:
Inclusion Criteria:

Acromegaly:

* Male or female patients ≥18 years of age
* Acromegaly currently treated with Sandostatin LAR

NET:

* Male or female patients ≥18 years of age
* Functional, well-differentiated (Grade 1 or Grade 2) NET with symptoms of carcinoid syndrome (number of bowel movements and/or flushing)
* Currently treated with Sandostatin LAR for symptom control

Exclusion Criteria:

Acromegaly:

* Inadequate bone marrow function
* Abnormal coagulation or chronic treatment with warfarin or coumarin derivates
* Impaired liver, cardiac and/or renal function
* Known gallbladder, bile duct disease or pancreatitis
* Diabetes with poorly controlled blood glucose levels despite adequate therapy
* Hypothyroidisms not adequately treated

NET:

* Poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, pancreatic islet cell carcinoma, insulinoma, glucagonoma, gastrinoma, goblet cell carcinoid, typical and atypical lung carcinoids, large cell neuroendocrine carcinoma and small cell carcinoma
* Carcinoid syndrome refractory to treatment with conventional doses of somatostatin analogues (SSAs)
* Inadequate bone marrow function
* Abnormal coagulation or chronic treatment with warfarin or coumarin derivates
* Impaired liver, cardiac and/or renal function
* Known gallbladder, bile duct disease or pancreatitis
* Short-bowel syndrome
* Diabetics with poorly controlled blood glucose levels despite adequate therapy
* Hypothyroidism, not adequately treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Pavel, Professor, Principal Investigator — Charité Campus Virchow Klinikum, Berlin, Germany
Locations (10):
- France (2):
  - Hospices Civils de Lyon, Bron
  - CHU Rouen, Hôpital Charles Nicolle, Rouen
- Germany (3):
  - Abteilung: Klinische Studien, Bad Berka
  - Charité Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Essen, Essen
- Italy (4):
  - RCCS Azienda Ospedaliera Universitaria San Martino IST, Genova
  - Fondazione Irccs Ca' Granda, Milan
  - Università degli Studi di Napoli Federico II, Napoli
  - Istituto Clinico Humanitas, Rozzano
- Akademiska sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Pavel M, Borson-Chazot F, Cailleux A, Horsch D, Lahner H, Pivonello R, Tauchmanova L, Darstein C, Olsson H, Tiberg F, Ferone D. Octreotide SC depot in patients with acromegaly and functioning neuroendocrine tumors: a phase 2, multicenter study. Cancer Chemother Pharmacol. 2019 Feb;83(2):375-385. doi: 10.1007/s00280-018-3734-1. Epub 2018 Dec 8. PMID 30535537

RESULTS

PARTICIPANT FLOW:
Groups:
- CAM2029 10 mg q2w (Acromegaly); CAM2029 10 mg q2w (NET): CAM2029 (octreotide FluidCrystal® injection depot) 10 mg, subcutaneous injection every two weeks
  octreotide FluidCrystal® injection depot
- CAM2029 20 mg q4w (Acromegaly); CAM2029 20 mg q4w (NET): CAM2029 (octreotide FluidCrystal® injection depot) 20 mg, subcutaneous injection once monthly
  octreotide FluidCrystal® injection depot
Period: Overall Study
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET)
Started | 3 | 4 | 1 | 4
Completed | 3 | 4 | 1 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET) | Total
Number analyzed (Participants) | 3 | 4 | 1 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 2 | 6
  >=65 years | 2 | 2 | 0 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14.93) | 62.5 (4.80) | 59 (0) | 64.8 (4.11) | 62.1 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 3
  Male | 2 | 2 | 1 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Italy | 2 | 1 | 0 | 0 | 3
  France | 1 | 3 | 0 | 1 | 5
  Germany | 0 | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) AUC
Description: Pharmacokinetics (PK) of octreotide after injection of Sandostatin Long-acting Release (LAR) was determined for the dosing period Day -28 to Day 0; AUC0-28d (day*ng/mL).
  AUC0-28d: AUC from 0 to 28 days over the final dosing interval (day*ng/mL) for Sandostatin LAR.
Time Frame: Pre-dose; study Day -28- to Day 0 (PK analysis:Sandostatin (LAR®) sampling time points: 0, 1hour, 24hours, 7days, 14days, 21days and 28days)
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: day*ng/mL
Groups:
- Sandostatin LAR 10 mg (Acromegaly); Sandostatin LAR 30mg (Acromegaly); Sandostatin LAR 20 mg (NET); Sandostatin LAR 30 mg (NET): Study injection (period 0) pre-CAM2029 treatment (day -28 to D0) of their ongoing maintenance therapy with Sandostatin LAR
Arm/Group | Sandostatin LAR 10 mg (Acromegaly) | Sandostatin LAR 30mg (Acromegaly) | Sandostatin LAR 20 mg (NET) | Sandostatin LAR 30 mg (NET)
Number analyzed (Participants) | 1 | 4 | 1 | 4
day*ng/mL | 6.23 (NA) — Single participant analyzed | 24.1 (11.6) | 27.8 (NA) — Single participant analyzed | 39.9 (20.5)

2. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) AUC.
Description: Pharmacokinetics (PK) of octreotide after administrations of CAM2029 was determined for the dosing period Day 0 to Day 84 ; AUC0-28d (day*ng/mL).
  AUC0-28d: AUC from 0 to 28 days over the dosing intervals (day*ng/mL) for CAM2029 20 mg q4w and CAM2029 10 mg q2w (to estimate AUC0-28d for those patients receiving CAM2029 10 mg q2w, AUC0-14d was multiplied by a factor of 2 as an estimate of the AUC0-28d) dosing intervals
Time Frame: (Day 0) to Day 84 (PK analysis:CAM2029 sampling time points: CAM2029 10mg q2w; 0, 2hours, 24hours, 48hours, 7days and 14days CAM2029 20mg q4w; 0, 2hours, 24hours, 48hours, 7days, 21days and 28days)
Population: Pharmacokinetic population, two patients excluded from the CAM2029 20mg Acromegaly due to incorrect dose.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET)
Number analyzed (Participants) | 3 | 2 | 1 | 4
day*ng/mL
  AUC0-28d (day*ng/mL) Day 0: number analyzed (Participants) | 3 | 2 | 1 | 3
  AUC0-28d (day*ng/mL) Day 0 | 92.9 (36.8) | 72.4 (6.73) | 72.9 (NA) — Single partcipant analyzed | 135 (37.8)
  AUC0-28d (day*ng/mL) Day 56: number analyzed (Participants) | 2 | 2 | 1 | 4
  AUC0-28d (day*ng/mL) Day 56 | 95.6 (63.3) | 78.5 (20.0) | 83.3 (NA) — Single partcipant analyzed | 135 (34.7)

3. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) Ctrough
Description: Pharmacokinetics (PK) of octreotide after injection of Sandostatin Long-acting Release (LAR) was determined for the dosing period Day -28 to Day 0; Ctrough (ng/mL).
  Ctrough; Concentration levels assessed prior to next injection for the final (Sandostatin LAR) dosing interval (ng/mL).
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sandostatin LAR 10 mg (Acromegaly) | Sandostatin LAR 30mg (Acromegaly) | Sandostatin LAR 20 mg (NET) | Sandostatin LAR 30 mg (NET)
Number analyzed (Participants) | 1 | 4 | 1 | 3
ng/mL | 0.225 (NA) — Single participant analyzed | 1.20 (0.647) | 0.901 (NA) — Single participant analyzed | 1.27 (0.480)

4. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) Cmax
Description: Pharmacokinetics (PK) of octreotide after injection of Sandostatin Long-acting Release (LAR) was determined for the dosing period Day -28 to Day 0; Cmax (ng/mL).
  Cmax (ng/mL): Maximum observed plasma concentration over the final (Sandostatin LAR) dosing interval (ng/mL)
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sandostatin LAR 10 mg (Acromegaly) | Sandostatin LAR 30mg (Acromegaly) | Sandostatin LAR 20 mg (NET) | Sandostatin LAR 30 mg (NET)
Number analyzed (Participants) | 1 | 4 | 1 | 4
ng/mL | 0.349 (NA) — Single participant analyzed | 1.41 (0.693) | 1.68 (NA) — Single participant analyzed | 2.48 (1.79)

5. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) Ctrough
Description: Pharmacokinetics (PK) of octreotide after administrations of CAM2029 was determined for the dosing period Day 0 to Day 84; Ctrough (ng/mL).
  Ctrough; Concentration levels assessed prior to next injection for CAM2029 20 mg q4w and CAM2029 10 mg q2w dosing intervals (ng/mL)
Time Frame: as for outcome 2
Population: Pharmacokinetic population, two patients excluded from the CAM2029 20mg Acromegaly due to incorrect dose.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET)
Number analyzed (Participants) | 3 | 2 | 1 | 4
ng/ml
  Ctrough (ng/mL) Day 0 | 1.32 (0.422) | 0.403 (0.342) | 1.80 (NA) — Single participant analyzed | 1.81 (0.817)
  Ctrough (ng(mL) Day 56 | 1.03 (0.223) | 1.01 (0.365) | 1.27 (NA) — Single participant analyzed | 1.73 (0.965)

6. Primary Outcome: Pharmacokinetic (PK) Profile of Octreotide After Each Injection of CAM2029 as Compared With Baseline PK for Sandostatin® Long-acting Release (LAR®) Cmax.
Description: Pharmacokinetics (PK) of octreotide after administrations of CAM2029 was determined for the dosing period Day 0 to Day 84 ; Cmax (ng/mL).
  Cmax (ng/mL): Maximum observed plasma concentration over CAM2029 20 mg q4w and CAM2029 10 mg q2w dosing intervals (ng/mL)
Time Frame: as for outcome 2
Population: Pharmacokinetic population, two patients excluded from the CAM2029 20mg Acromegaly due to incorrect dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET)
Number analyzed (Participants) | 3 | 2 | 1 | 4
ng/mL
  Cmax (ng/mL) Day 0: number analyzed (Participants) | 3 | 2 | 1 | 3
  Cmax (ng/mL) Day 0 | 10.4 (6.62) | 13.4 (4.31) | 6.33 (NA) — Single participant analyzed | 16.3 (8.67)
  Cmax (ng/mL) Day 56: number analyzed (Participants) | 2 | 2 | 1 | 4
  Cmax (ng/mL) Day 56 | 10.6 (10.2) | 11.3 (2.58) | 5.61 (NA) — Single participant analyzed | 15.7 (4.05)

7. Secondary Outcome: Number of Adverse Events and Serious Adverse Events
Description: Safety (number of adverse events and serious adverse events) after repeated doses of CAM2029 (assessment period from Day 0 to Day 84) and single dose Sandostatin LAR (assessment period Day -28 to Day 0)
Time Frame: Day -28 to Day 84
Population: Safety population (n=12). Patients treated with Sandostatin LAR Day -28 to 0 and CAM2029 (Day 0 to Day 84)
Measure: Count of Participants; unit: Participants
Groups:
- Sandostatin LAR (Acromegaly): Period day -28 to day 0 All acromegaly patients and all treatment groups
- Sandostain LAR (NET): Period day-28 to 0 All NET patient and all treatment groups
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET) | Sandostatin LAR (Acromegaly) | Sandostain LAR (NET)
Number analyzed (Participants) | 3 | 4 | 1 | 4 | 7 | 5
Participants | 2 | 4 | 0 | 2 | 4 | 2

8. Secondary Outcome: CAM2029 Effect on Insulin-like Growth Factor (IGF-1) (Acromegaly)
Description: Data is presented as number of patients
  * Within the reference limits (see below)
  * Above ULN (Upper Limits of Normal)
  In the Acromegaly group both males and females were included the age was between 42-70 years. The IGF normal range for the different genders and age are presented below.
  REFERENCE VALUES
  Males (NMOL/L) 8.34-27.44 (41-45 years) 7.7-26.36 (46-50 years) 7.3-26.34 (51-55 years) 6.64-25.44 (56-60 years) 6.17-25.02 (61-65 years) 5.96-25.48 (66-70 years)
  Females (NMOL/L) 8.06-26.89 (41-45 years) 7.39-25.44 (46-50 years) 6.92-24.98 (51-55 years) 5.92-22.7 (56-60 years) 5.42-21.96 (61-65 years) 5.07-21.97 (66-70 years)
Time Frame: Day 84
Population: Pharmacokinetic population (5 acromegaly subjects total)
Measure: Number; unit: participants
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly)
Number analyzed (Participants) | 3 | 2
participants
  Within Normal Limits | 2 | 1
  Above ULN | 1 | 1

9. Secondary Outcome: CAM2029 Effect on Growth Hormone (GH) (Acromegaly)
Description: GH (growth hormone) levels measured on Day 84 in patients with acromegaly
Time Frame: Day 84
Population: Pharmacokinetic population (5 acromegaly patients)
Measure: Number; unit: participants
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acromegaly)
Number analyzed (Participants) | 3 | 2
participants
  GH level < 2.5 μg/L | 2 | 2
  GH level >2.5 μg/L | 1 | 0

10. Other Pre Specified Outcome: To Assess the Symptoms of Carcinoid Syndrome (Number of Bowel Movements and Flushing) and the Use of Rescue Medication Versus Baseline (by Using Patient Diaries) (NET)
Description: Number of bowel movements and flushing during period 0 and 1, data is presented as patients experience symptoms
  Bowel movement without flushing Bowel movement and flushing No Bowel movement or Flushing
Time Frame: Baseline (Day 0), Day 84
Population: Pharmacokinetic population
Measure: Number; unit: participants
Arm/Group | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET)
Number analyzed (Participants) | 1 | 4
participants
  Bowel movements without flushing | 1 | 0
  Bowel movements with flushing | 0 | 2
  No Bowel movement or Flushing | 0 | 2

ADVERSE EVENTS:
Groups:
- CAM2029 10 mg q2w (Acromegaly); CAM2029 10 mg q2w (NET): CAM2029 (octreotide FluidCrystal® injection depot) 10 mg, subcutaneous injection every two weeks
  octreotide FluidCrystal® injection depot Day 0-84
- CAM2029 20 mg q4w (Acormegaly); CAM2029 20 mg q4w (NET): CAM2029 (octreotide FluidCrystal® injection depot) 20 mg, subcutaneous injection once monthly
  octreotide FluidCrystal® injection depot Day 0-84
- Sandostatin LAR (Acromegaly): Sandostatin LAR Day-28 to day 0 All acromegaly patients, all treatment groups
- Sandostatin LAR (NET): Sandostatin LAR Day -28 to day 0 All NET patients, all treatment groups
Arm/Group | CAM2029 10 mg q2w (Acromegaly) | CAM2029 20 mg q4w (Acormegaly) | CAM2029 10 mg q2w (NET) | CAM2029 20 mg q4w (NET) | Sandostatin LAR (Acromegaly) | Sandostatin LAR (NET)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 1/4 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 0/1 | 2/4 | 4/7 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2029 10 mg q2w (Acromegaly) (N=3) | CAM2029 20 mg q4w (Acormegaly) (N=4) | CAM2029 10 mg q2w (NET) (N=1) | CAM2029 20 mg q4w (NET) (N=4) | Sandostatin LAR (Acromegaly) (N=7) | Sandostatin LAR (NET) (N=5)
Anastomotic ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — D39, patient noticed intermittent episodes of blood in stools due to a ulceration of a previous anastomosis. Patient received the last injection dose D57 and was hospitalized for investigations of bleeding, resolved on D60, not related to treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2029 10 mg q2w (Acromegaly) (N=3) | CAM2029 20 mg q4w (Acormegaly) (N=4) | CAM2029 10 mg q2w (NET) (N=1) | CAM2029 20 mg q4w (NET) (N=4) | Sandostatin LAR (Acromegaly) (N=7) | Sandostatin LAR (NET) (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetitie (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insulin like growth factor increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less